CLINICAL TRIAL: NCT02388607
Title: Sustained Attention Abilities, Attentional Resources and Cognitive Control Mechanisms in Schizophrenia
Brief Title: Sustained Attention Abilities in Schizophrenia
Acronym: ACCRAS
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Other Study IDs: 5972
Record Dates: First submitted 2014-12-10; First posted 2015-03-17 (Estimated); Last update posted 2021-09-14 (Actual); Status verified 2021-09

CONDITIONS: Schizophrenic Psychoses
MeSH Terms: interventions — Weights and Measures

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- assessing attention span: * Electrophysiological measurements (evocated potentials and spectral densities)
  * Clinical scales and subjective assessments of difficulty of the tasks performed, and commitment to the task
  Interventions: Other: measurements

INTERVENTIONS:
Other: measurements — performance measurements

SUMMARY:
Schizophrenia is a psychiatric pathology, which concerns around 1% of adult population. It is characterized by clinical symptoms combining positive and negative symptoms and thinking disorganization. Schizophrenia is also characterized by cognitive deficits, likely to play an important part in adaptation of these patients in their every-day life, and to affect their clinical symptomatology. Among them, there are deficits in sustained attention which are associated with a difficulty for these patients to maintain efficiently their cognitive activity on a source of stimulation or task. This basic attentional process is fundamental for the efficiency of the overall of cognitive processes, and so for all behaviors directed on an aim. The question of whether or not patients with schizophrenia have difficulty sustaining attention is of high relevance, in the sense that it could undermine performance on nearly any task and so provide a compelling causal explanation of many other impairments observed in these patients. Yet it has not been conclusively answered in over four decades of research. Consequently, the main objective of the protocol is to evaluate sustained attention abilities in schizophrenic patients and to better understand the specific functioning of cognitive and neural mechanisms underlying these abilities (attentional resources and cognitive control mechanisms).

ELIGIBILITY:
Inclusion Criteria:

* age between 18 and 60 years (include)
* men or women volunteers, hospitalized or not
* subject affiliated to an health insurance
* subject having signed an informed consent (for patients):
* presence of DSM-IV TR criteria for schizophrenia (American Psychiatric Association, 1994)

Exclusion criteria

* a major somatic disorder or non stabilized
* medical history likely to affect cerebral anatomy or to be linked to an abnormality (neonatal distress, neurochirurgical intervention, neurological disorders, stroke attack)
* any disorders involved in the use of a psycho-active substance (as defined by the DSM-IV)
* sensory disabling impairments, and specifically visual acuity < 8
* general anaesthesia during the 3 months before the study
* pregnancy (declared by the subject)
* persons in an emergency situation
* persons deprived in any way of their liberty
* persons in period of exclusion in an other protocol
* use of psychotropic substance during the 3 weeks before the study
* use of benzodiazepines

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: 40 schizophrenic patients versus 40 healthy subjects matched
Sampling Method: Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2015-03 (Actual); Primary Completion 2023-03 (Estimated); Study Completion 2023-03 (Estimated)

PRIMARY OUTCOMES:
Assess sustained attention span of patients with schizophrenia | two half-days
  Subjects are involved in 4 different attentional tasks during which behavioral and electrophysiological measures are recorded in order to evaluate sustained attention abilities and the specific functioning of cognitive and neural mechanisms underlying these abilities in schizophrenic patients.

SECONDARY OUTCOMES:
Study the specific mechanisms underlying attention skills supported in schizophrenic patients | two half-days
  Subjects are involved in 4 different attentional tasks during which behavioral and electrophysiological measures are recorded in order to evaluate sustained attention abilities and the specific functioning of cognitive and neural mechanisms underlying these abilities in schizophrenic patients.

CONTACTS AND LOCATIONS:
Overall Officials: Giersch Anne, MD, Principal Investigator — Les Hôpitaux Universitaires de Strasbourg; Bonnefond Anne, PHD, Study Chair — Institut National de la Santé Et de la Recherche Médicale, France
Locations (1):
- Service de psychiatrie, Strasbourg, France